CLINICAL TRIAL: NCT00515008
Title: Tai Chi Mind-Body Therapy for Fibromyalgia: a Pilot Single-Blind Randomized Controlled Trial.
Brief Title: Tai Chi Mind-Body Therapy for Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); American College of Rheumatology Research and Education Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21AT003621 (NIH); R21AT003621 (NIH)
Record Dates: First submitted 2007-08-09; First posted 2007-08-13 (Estimated); Results first posted 2016-03-08 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-02

CONDITIONS: Fibromyalgia
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tai Chi Intervention (Experimental): The tai chi intervention took place twice a week for 12 weeks, and each session lasted for 60 minutes. Classes were taught by a tai chi master with more than 20 years of teaching experience. In the first session, he explained the theory behind tai chi and its procedures and provided participants with printed materials on its principles and techniques. In subsequent sessions, participants practiced 10 forms from the classic Yang style of tai chi 18 under his instruction. Each session included a warm-up and self-massage, followed by a review of principles, movements, breathing techniques, and relaxation in tai chi. Throughout the intervention period, participants were instructed to practice tai chi at home for at least 20 minutes each day. At the end of the 12-week intervention, participants were encouraged to maintain their tai chi practice, using an instructional DVD, up until the follow-up visit at 24 weeks.
  Interventions: Behavioral: Tai Chi Intervention
- Control Intervention (Placebo Comparator): Our wellness education and stretching program similarly included 60-minute sessions held twice a week for 12 weeks.19 At each session, a variety of health professionals provided a 40-minute didactic lesson on a topic relating to fibromyalgia, including the diagnostic criteria; coping strategies and problem-solving techniques; diet and nutrition; sleep disorders and fibromyalgia; pain management, therapies, and medications; physical and mental health; exercise; and wellness and lifestyle management.20 For the final 20 minutes of each class, participants practiced stretching exercises supervised by the research staff. Stretches involved the upper body, trunk, and lower body and were held for 15 to 20 seconds. Participants were instructed to practice stretching at home for 20 minutes a day.
  Interventions: Behavioral: Control Intervention

INTERVENTIONS:
Behavioral: Tai Chi Intervention — The tai chi intervention took place twice a week for 12 weeks, and each session lasted for 60 minutes. Classes were taught by a tai chi master with more than 20 years of teaching experience. In the first session, he explained the theory behind tai chi and its procedures and provided participants with printed materials on its principles and techniques. In subsequent sessions, participants practiced 10 forms from the classic Yang style of tai chi18 under his instruction. Each session included a warm-up and self-massage, followed by a review of principles, movements, breathing techniques, and relaxation in tai chi. Throughout the intervention period, participants were instructed to practice tai chi at home for at least 20 minutes each day. At the end of the 12-week intervention, participants were encouraged to maintain their tai chi practice, using an instructional DVD, up until the follow-up visit at 24 weeks.
  Arms: Tai Chi Intervention
Behavioral: Control Intervention — Our wellness education and stretching program similarly included 60-minute sessions held twice a week for 12 weeks.19 At each session, a variety of health professionals provided a 40-minute didactic lesson on a topic relating to fibromyalgia, including the diagnostic criteria; coping strategies and problem-solving techniques; diet and nutrition; sleep disorders and fibromyalgia; pain management, therapies, and medications; physical and mental health; exercise; and wellness and lifestyle management.20 For the final 20 minutes of each class, participants practiced stretching exercises supervised by the research staff. Stretches involved the upper body, trunk, and lower body and were held for 15 to 20 seconds. Participants were instructed to practice stretching at home for 20 minutes a day.
  Arms: Control Intervention

SUMMARY:
The purpose of this study is to obtain preliminary data on the effects of Tai Chi on musculoskeletal pain, fatigue, sleep quality, psychological distress, physical performance,and health status in 60 patients with fibromyalgia.

DETAILED DESCRIPTION:
Fibromyalgia (FM) is a common, complex chronic condition marked by diffuse musculoskeletal pain, fatigue, functional impairment, disability, and psychological distress that affects 6-10 million people in the United States (US). There are currently no satisfactory pharmacological or non-pharmacological treatments for FM. New cost-effective strategies that reduce musculoskeletal pain and improve emotional and physical functioning as well as quality of life in people with FM are urgently needed.

Tai Chi is a traditional Chinese discipline with both physical and mental components that appears to benefit a variety of chronic conditions. The physical component provides exercise that is consistent with that recommended for FM (muscle conditioning and aerobic cardiovascular exercise), while the mental component has the potential to improve psychological well-being. These effects are especially pertinent for the treatment of individuals with FM.

This is a pilot randomized controlled trial of Tai Chi for fibromyalgia. We plan to enroll 60 patients with fibromyalgia over a two year period. Participants are randomized to either a Tai Chi program or an attention control intervention. Assessments are performed at baseline, week 12 and week 24. This study will provide preliminary data on the potential acceptability and safety of Tai Chi for FM and will help guide the design of a future large-scale study of the efficacy of this alternative therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or older
* Fulfills the American College of Rheumatology (ACR) 1990 diagnostic criteria for FM. (1) a history of widespread musculoskeletal pain on the right and left sides of the body as well as above and below the waist for a minimum duration of 3 months, and (2) pain in 11 or more of 18 specific tender points with moderate or greater tenderness reported upon digital palpation.
* Physically able to participate in both the Tai Chi and stretching and education programs according to their primary care physician.
* Willing to complete the 12-week study, including twice-a-week Tai Chi or stretching and education sessions

Exclusion Criteria

* Prior experience with Tai Chi or other similar types of Complementary and Alternative Medicine in the past 6 months such as Qi gong and yoga since these share some of the principles of Tai Chi
* Any health condition limiting the ability to participate as determined by a primary care physician
* Any other diagnosed medical condition that is known to contribute to FM symptomatology that is not under adequate control or cannot be expected to remain under adequate control for the study period such as thyroid disease, inflammatory arthritis, scleroderma, systemic lupus erythematosus, systemic sclerosis, rheumatoid arthritis, myositis and vasculitis or Sjogren's syndrome
* Not English-Speaking
* Positive pregnancy test or planning pregnancy within the study period
* Inability to pass the Mini-Mental Status examination (score below 24)
* Enrollment in any other clinical trial within the last 30 days
* Plan to permanently relocate from the region during the trial period

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chenchen Wang, MD, MSc, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Division of Rheumatology, Boston, Massachusetts, United States

REFERENCES:
- [Background] Wang C, Collet JP, Lau J. The effect of Tai Chi on health outcomes in patients with chronic conditions: a systematic review. Arch Intern Med. 2004 Mar 8;164(5):493-501. doi: 10.1001/archinte.164.5.493. PMID 15006825
- [Background] Wang C, Roubenoff R, Lau J, Kalish R, Schmid CH, Tighiouart H, Rones R, Hibberd PL. Effect of Tai Chi in adults with rheumatoid arthritis. Rheumatology (Oxford). 2005 May;44(5):685-7. doi: 10.1093/rheumatology/keh572. Epub 2005 Mar 1. No abstract available. PMID 15741197
- [Background] Wang C. Tai Chi improves pain and functional status in adults with rheumatoid arthritis: results of a pilot single-blinded randomized controlled trial. Med Sport Sci. 2008;52:218-229. doi: 10.1159/000134302. PMID 18487901
- [Derived] Wang C, Schmid CH, Rones R, Kalish R, Yinh J, Goldenberg DL, Lee Y, McAlindon T. A randomized trial of tai chi for fibromyalgia. N Engl J Med. 2010 Aug 19;363(8):743-54. doi: 10.1056/NEJMoa0912611. PMID 20818876

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We conducted the trial from July 2007 through May 2009 at Tufts Medical Center, a tertiary care academic hospital in Boston.
Pre-assignment Details: 90 Underwent baseline evaluation. 24 Were excluded:
  1 Did not have fibromyalgia 4 Were physically unable to participate 17 Had scheduling conflicts
  1 Was currently practicing tai chi
  1 Had preexisting medical condition
Groups:
- Tai Chi Group: 12-week Tai Chi Program.: The tai chi intervention took place twice a week for 12 weeks, and each session lasted for 60 minutes. Classes were taught by a tai chi master with more than 20 years of teaching experience. In the first session, he explained the theory behind tai chi and its procedures and provided participants with printed materials on its principles and techniques. In subsequent sessions, participants practiced 10 forms from the classic Yang style of tai chi under his instruction. Each session included a warm-up and self-massage, followed by a review of principles, movements, breathing techniques, and relaxation in tai chi. Throughout the intervention period, participants were instructed to practice tai chi at home for at least 20 minutes each day. At the end of the 12-week intervention, participants were encouraged to maintain their tai chi practice, using an instructional DVD, up until the follow-up visit at 24 weeks.
- Control Group: 12-week Stretching and Wellness Education Program: Non-TC informational program. Our wellness education and stretching program similarly included 60-minute sessions held twice a week for 12 weeks. At each session, a variety of health professionals provided a 40-minute didactic lesson on a topic relating to fibromyalgia, including the diagnostic criteria; coping strategies and problem-solving techniques; diet and nutrition; sleep disorders and fibromyalgia; pain management, therapies, and medications; physical and mental health; exercise; and wellness and lifestyle management. For the final 20 minutes of each class, participants practiced stretching exercises supervised by the research staff. Stretches involved the upper body, trunk, and lower body and were held for 15 to 20 seconds. Participants were instructed to practice stretching at home for 20 minutes a day.
Period: Overall Study
Arm/Group | Tai Chi Group | Control Group
Started | 33 | 33
Completed 12 Week Evaluation | 32 | 29
Completed | 30 | 29
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 1 | 0
Not completed — Declined | 0 | 3
Not completed — Left the Boston Area | 1 | 1
Not completed — Scheduling conflict | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Tai Chi Group: 12-week Tai Chi Program.: 12-week Tai Chi classes
- Control Group: 12-week Stretching and Wellness Education Program: Non-TC informational program
- Total: Total of all reporting groups
Arm/Group | Tai Chi Group | Control Group | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (11.8) | 50.5 (10.5) | 50 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 29 | 57
  Male | 5 | 4 | 9
Region of Enrollment [Number; unit: participants]
  United States | 33 | 33 | 66
FIQ score [Mean (Standard Deviation); unit: units on a scale] — Fibromyalgia Impact Questionnaire (FIQ) is a well-validated, multidimensional measure of the overall severity of fibromyalgia as rated by patients. Categories include the intensity of pain, physical functioning, fatigue, morning tiredness, stiffness, depression, anxiety, job difficulty, and overall well-being.21 The total score ranges from 0 to 100, with higher scores indicating more severe symptoms.
  units on a scale | 62.9 (15.5) | 68 (11) | 65.5 (13.3)
Patient's global assessment score [Mean (Standard Deviation); unit: units on a scale] — Patients' global assessment score was assessed separately by the participant, who was unaware of the group assignment, with the use of a visual-analogue scale (VAS) (range, 0 to 10,with higher scores indicating greater pain).
  units on a scale | 5.8 (2.3) | 6.3 (1.8) | 6.1 (2.1)
Physician's global assessment score [Mean (Standard Deviation); unit: units on a scale] — Physicians' global assessment score was assessed separately by the study physician, who was unaware of the group assignment, with the use of a visual-analogue scale (VAS) (range, 0 to 10,with higher scores indicating greater pain).
  units on a scale | 5.7 (1.9) | 5.6 (2.4) | 5.7 (2.2)
PSQI score [Mean (Standard Deviation); unit: units on a scale] — The Pittsburgh Sleep Quality Index (PSQI) is a self-report measure of sleep quality(range, 0 to 21, with higher scores indicating worse sleep quality)
  units on a scale | 13.9 (3.1) | 13.5 (3.7) | 13.7 (3.4)
6-Minute walk test [Mean (Standard Deviation); unit: yards] | 522.1 (102.7) | 501.2 (106.6) | 511.7 (104.7)
Body-mass index [Mean (Standard Deviation); unit: kg/m^2] | 33.9 (8.9) | 31.5 (7.4) | 32.7 (8.2)
SF-36 score- Physical component [Mean (Standard Deviation); unit: units on a scale] — The Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) Physical Component is the summary score for the physical quality-of-life components (range, 0 to 100, with higher scores indicating better health status)
  units on a scale | 28.5 (8.4) | 28.0 (7.8) | 28.3 (8.1)
SF-36 score- Mental component [Mean (Standard Deviation); unit: units on a scale] — The Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) Mental Component is the summary score for the mental quality-of-life components (range, 0 to 100, with higher scores indicating better health status)
  units on a scale | 42.6 (12.2) | 37.8 (10.5) | 40.2 (11.4)
CES-D score [Mean (Standard Deviation); unit: units on a scale] — The Center for Epidemiologic Studies (CES-D) Depression Scale (range, 0 to 60, with higher scores indicating more severe depression), is a self-report measure of depressive symptoms.
  units on a scale | 22.6 (9.2) | 27.8 (9.2) | 25.2 (9.2)
CPSS score [Mean (Standard Deviation); unit: units on a scale] — The Chronic Pain Self-Efficacy Scale (CPSS) is a self-report score measuring self-efficacy with respect to chronic pain (range, 1 to 10, with higher scores indicating greater self-efficacy).
  units on a scale | 5.2 (1.9) | 4.6 (2.2) | 4.9 (2.1)
Outcome Expectations for Exercise score [Mean (Standard Deviation); unit: units on a scale] — The Outcome Expectations for Exercise Scale (range, 1 to 5, with 1 indicating no expectations for exercise and 5 the highest expectations for exercise) is a self-report measure of outcome expectations for exercise.
  units on a scale | 3.7 (0.8) | 3.9 (0.7) | 3.8 (0.8)
High School or Higher Education [Number; unit: participants] | 31 | 30 | 61
Duration of fibromyalgia-related pain - yr [Mean (Standard Deviation); unit: years] | 11.8 (6.9) | 10.0 (7.2) | 10.9 (7.1)
White race [Number; unit: participants] | 20 | 17 | 37

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline of Fibromyalgia Impact Questionnaire Score
Description: Fibromyalgia Impact Questionnaire (FIQ) is a well-validated, multidimensional measure of the overall severity of fibromyalgia as rated by patients. Categories include the intensity of pain, physical functioning, fatigue, morning tiredness, stiffness, depression, anxiety, job difficulty, and overall well-being.21 The total score ranges from 0 to 100, with higher scores indicating more severe symptoms.
Time Frame: wks 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Tai Chi: The tai chi intervention took place twice a week for 12 weeks, and each session lasted for 60 min- utes. Classes were taught by a tai chi master with more than 20 years of teaching experience. In the first session, he explained the theory behind tai
  chi and its procedures and provided participants with printed materials on its principles and tech- niques. In subsequent sessions, participants prac- ticed 10 forms from the classic Yang style of tai chi18 under his instruction. Each session included a warm-up and self-massage, followed by a review of principles, movements, breathing techniques, and relaxation in tai chi. Throughout the inter- vention period, participants were instructed to practice tai chi at home for at least 20 minutes each day. At the end of the 12-week intervention, participants were encouraged to maintain their tai chi practice, using an instructional DVD, up until the follow-up visit at 24 weeks.
- Control Group: Our wellness education and stretching program similarly included 60-minute sessions held twice a week for 12 weeks.19 At each session, a variety of health professionals provided a 40-minute didactic lesson on a topic relating to fibromyal- gia, including the diagnostic criteria; coping strat- egies and problem-solving techniques; diet and nutrition; sleep disorders and fibromyalgia; pain management, therapies, and medications; physi- cal and mental health; exercise; and wellness and
  lifestyle management.20 For the final 20 minutes of each class, participants practiced stretching ex- ercises supervised by the research staff. Stretches involved the upper body, trunk, and lower body and were held for 15 to 20 seconds. Participants were instructed to practice stretching at home for 20 minutes a day.
Arm/Group | Tai Chi | Control Group
Number analyzed (Participants) | 33 | 33
units on a scale | -27.8 [-33.8 to -21.8] | -9.4 [-15.5 to -3.4]

2. Secondary Outcome: Mean Change From Baseline of VAS Physicians' Global Assessment of Fibromyalgia Severity
Description: Physicians' global assessment score was assessed separately by the study physician, who was unaware of the group assignment, with the use of a visual-analogue scale (VAS) (range, 0 to 10,with higher scores indicating greater pain).
Time Frame: Wks 12
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tai Chi | Control Group
Number analyzed (Participants) | 33 | 33
units on a scale | -1.0 [-1.7 to -0.4] | 0.02 [-0.6 to 0.7]

3. Secondary Outcome: Mean Change From Baseline of Patient's Global Assessment Score
Description: Patients' global assessment score was assessed separately by the participant, who was unaware of the group assignment, with the use of a visual-analogue scale (VAS) (range, 0 to 10,with higher scores indicating greater pain).
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tai Chi | Control Group
Number analyzed (Participants) | 33 | 33
units on a scale | -2.5 [-3.3 to -1.7] | -0.6 [-1.4 to 0.2]

4. Secondary Outcome: Mean Change From Baseline PSQI Score
Description: The Pittsburgh Sleep Quality Index (PSQI) is a self-report measure of sleep quality(range, 0 to 21, with higher scores indicating worse sleep quality)
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tai Chi Group | Control Group
Number analyzed (Participants) | 33 | 33
units on a scale | -3.6 [-4.8 to -2.4] | -0.7 [-1.9 to 0.5]

5. Secondary Outcome: Mean Change From Baseline of 6-Minute Walk Test
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: yards
Arm/Group | Tai Chi Group | Control Group
Number analyzed (Participants) | 33 | 33
yards | 60.6 [37.9 to 83.3] | 16.3 [-6.4 to 38.9]

6. Secondary Outcome: Mean Change From Baseline SF-36 Score Physical Component
Description: The Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) Physical Component is the summary score for the physical quality-of-life components (range, 0 to 100, with higher scores indicating better health status)
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tai Chi Group | Control Group
Number analyzed (Participants) | 33 | 33
units on a scale | 8.5 [5.7 to 11.3] | 1.4 [-1.5 to 4.2]

7. Secondary Outcome: Mean Change From Baseline SF-36 Score Mental Component
Description: The Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) Mental Component is the summary score for the mental quality-of-life components (range, 0 to 100, with higher scores indicating better health status)
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tai Chi Group | Control Group
Number analyzed (Participants) | 33 | 33
units on a scale | 7.7 [3.9 to 11.6] | 6.1 [0.7 to 11.6]

8. Secondary Outcome: Mean Change From Baseline CES-D Score
Description: The Center for Epidemiologic Studies (CES-D) Depression Scale (range, 0 to 60, with higher scores indicating more severe depression), is a self-report measure of depressive symptoms.
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tai Chi Group | Control Group
Number analyzed (Participants) | 33 | 33
units on a scale | -8.1 [-10.9 to -5.3] | -2.3 [-5.1 to 0.6]

9. Secondary Outcome: Mean Change From Baseline CPSS Score
Description: The Chronic Pain Self-Efficacy Scale (CPSS) is a self-report score measuring self-efficacy with respect to chronic pain (range, 1 to 10, with higher scores indicating greater self-efficacy).
Time Frame: 12 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tai Chi Group | Control Group
Number analyzed (Participants) | 33 | 33
units on a scale | 1.5 [0.7 to 2.2] | 0.5 [-0.3 to 1.2]

ADVERSE EVENTS:
Time Frame: 24 months
Description: We monitored adverse events, using a standard case report form at each visit. This form included a description of all unanticipated benefits and undesirable experiences, particularly falls and exacerbations of fibromyalgia symptoms.
Arm/Group | Tai Chi Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/33
Other Adverse Events (participants affected / at risk) | 0/33 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No